CLINICAL TRIAL: NCT00225849
Title: Japanese Primary Prevention Project With Aspirin in the Elderly With One or More Risk Factors of Vascular Events: JPPP
Brief Title: Japanese Primary Prevention Project With Aspirin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Health, Labour and Welfare, Japan (Other Government)
Collaborators: Japan Heart Foundation (Other); Bayer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JPPP-05-07; MHLW2004-CV(Adult disease)-010
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2005-09-26 (Estimated); Status verified 2005-09

CONDITIONS: Hypertension; Hyperlipidemia; Diabetes Mellitus
Keywords: Aspirin; Primary prevention
MeSH Terms: conditions — Hypertension; Hyperlipidemias; Diabetes Mellitus | interventions — Aspirin

INTERVENTIONS:
Drug: Aspirin

SUMMARY:
The purpose of this study is to investigate the balance between the risks and benefits of primary prevention by Aspirin in elderly Japanese patients with one or more cerebro/cardiovascular risk factors

DETAILED DESCRIPTION:
Cerebro/cardiovascular (CV) death accounts for approximately 30% of total deaths in Japan and therefore it is important to establish a preventive treatment for CV events from the point of public health. The guidelines proposed by a joint study group centering on the Japanese Circulation Society, recommend administration of aspirin to patients with multiple risk factors for primary prevention of arteriosclerotic diseases. In addition, the 2002 AHA guidelines recommend use of aspirin in patients with a 10% or higher 10-year risk of CV events. However, these descriptions are founded on randomized, comparative study results and epidemiological data obtained outside Japan, while no epidemiological data are available in Japan that would allow prediction and selection of patients who could benefit from primary prevention with aspirin. Although the benefit of aspirin for secondary prevention has been proven in Japanese patients, the benefits of primary prevention are still controversial.

JPPP is a multicenter, open-label, centrally randomized, controlled trial. In total, 10,000 elderly patients with one or more CV risk factors (age 60-85 years combined with hypertension, hyperlipidemia, and/or diabetes) will be assigned to enteric-coated aspirin (100mg/day) or control. The primary endpoint is composite event of CV death, nonfatal stroke (of any cause) and nonfatal myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients not previously diagnosed to have any arteriosclerotic disease, including coronary artery disease or cerebrovascular disease, but meeting any one or more of the following criteria (or on medication for any one or more of the following conditions).

  * Hypertension: SBP ≥ 140 mmHg or DBP ≥ 90 mmHg
  * Hyperlipidemia: Hypercholesterolemia (total cholesterol ≥ 220 mg/dL or LDL cholesterol ≥ 140 mg/dL) or Hypertriglyceridemia (Triglycerides ≥ 150 mg/dL) or Low-HDL cholesterolemia (HDL cholesterol < 40 mg/dL)
  * Diabetes: Fasting morning blood glucose ≥ 126 mg/dL or casual blood glucose ≥ 200 mg/dL or blood glucose at 2 hrs in the 75-g glucose tolerance test ≥ 200 mg/dL, or HbA1c ≥ 6.5%
* Age: 60 to 85 years
* Patients who can give written consent for participation in the study

Exclusion Criteria:

* Patients with a history of coronary artery disease or cerebrovascular disease (including transient ischemic attack)
* Patients with arteriosclerotic disease requiring surgery or intervention
* Patients who have or may have atrial fibrillation
* Patients being treated with aspirin, other antiplatelet agents or anticoagulants
* Patients using NSAIDs chronically
* Patients with a history of hypersensitivity to aspirin or salicylic acid
* Patients with peptic ulcers
* Patients with a bleeding tendency
* Patients with serious blood abnormalities
* Patients with aspirin-sensitive asthma or a history of the same
* Patients who are otherwise judged by the investigator to be unsuitable for enrollment in the study.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000
Dates: Start 2005-03; Study Completion 2010-09

PRIMARY OUTCOMES:
Composite event of cerebro/cardiovascular (CV) death, nonfatal cerebral stroke (of any cause) and nonfatal myocardial infarction (MI)

SECONDARY OUTCOMES:
CV death
Non CV death
Nonfatal cerebral stroke
Nonfatal MI
Angina pectoris
Transient ischemic attack
Arteriosclerotic disease requiring surgery or intervention
Extracranial bleeding requiring transfusion or admission
Severe side-effects that lead to interruption of the study medication.

CONTACTS AND LOCATIONS:
Overall Officials: Yasuo Ikeda, MD, Principal Investigator — Keio University
Locations (1):
- Keio University School of Medicine, Tokyo, Tokyo, Japan

REFERENCES:
- [Derived] Sugawara M, Goto Y, Yamazaki T, Teramoto T, Oikawa S, Shimada K, Uchiyama S, Ando K, Ishizuka N, Murata M, Yokoyama K, Uemura Y, Ikeda Y; Japanese Primary Prevention Project (JPPP) Study Group. Low-Dose Aspirin for Primary Prevention of Cardiovascular Events in Elderly Japanese Patients with Atherosclerotic Risk Factors: Subanalysis of a Randomized Clinical Trial (JPPP-70). Am J Cardiovasc Drugs. 2019 Jun;19(3):299-311. doi: 10.1007/s40256-018-0313-0. PMID 30565155
- [Derived] Uchiyama S, Ishizuka N, Shimada K, Teramoto T, Yamazaki T, Oikawa S, Sugawara M, Ando K, Murata M, Yokoyama K, Minematsu K, Matsumoto M, Ikeda Y; JPPP Study Group. Aspirin for Stroke Prevention in Elderly Patients With Vascular Risk Factors: Japanese Primary Prevention Project. Stroke. 2016 Jun;47(6):1605-11. doi: 10.1161/STROKEAHA.115.012461. Epub 2016 May 10. PMID 27165949
- [Derived] Ikeda Y, Shimada K, Teramoto T, Uchiyama S, Yamazaki T, Oikawa S, Sugawara M, Ando K, Murata M, Yokoyama K, Ishizuka N. Low-dose aspirin for primary prevention of cardiovascular events in Japanese patients 60 years or older with atherosclerotic risk factors: a randomized clinical trial. JAMA. 2014 Dec 17;312(23):2510-20. doi: 10.1001/jama.2014.15690. PMID 25401325